CLINICAL TRIAL: NCT06312618
Title: Efficacy of Propofol Versus Dexmedetomidine To Prevent Emergence Agitation After Sevoflurane Anesthesia In Children Undergoing Squint Surgery
Brief Title: Propofol Versus Dexmedetomidine Effect on Prevention Emergence Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MD292/2023
Record Dates: First submitted 2024-02-23; First posted 2024-03-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-02

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Propofol group (Active Comparator): children will be randomized to receive propofol 1mg/kg over 10 minutes
  Interventions: Drug: Propofol
- Group 2: Dexmedetomidine group (Active Comparator): children will be randomized to receive dexmedetomidine 0.2 mcg/kg over 10 minutes
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — After completion of the procedure and after regain muscle power sevoflurane administration will be ceased. children will be randomized to receive propofol
  1mg/kg over 10 minutes (group 1) .
  Other Names: Diprivan
  Arms: Group 1: Propofol group
Drug: Dexmedetomidine — After completion of the procedure and after regain muscle power sevoflurane administration will be ceased. children will be randomized to receive dexmedetomidine 0.2 mcg/kg over 10 minutes (group 2).
  Other Names: Precedex
  Arms: Group 2: Dexmedetomidine group

SUMMARY:
The goal of this clinical trial is to compare Propofol versus Dexmedetomidine in children undergoing squint surgery. The main question it aims to answer is:

• Which drug is more effective in preventing the appearance of Emergence Agitation in children after sevoflurane anesthesia in squint surgery, propofol or dexmedetomidine?

Emergence agitation (EA) is a period of restlessness, agitation, inconsolable crying, disorientation, delusions, and hallucinations with impaired cognition and memory that commonly occurs in children undergoing ophthalmic surgery especially after Short acting volatile agents such as sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients from 3 to 7 years.
* American Society of Anesthesiologists (ASA) Physical Status Class-I and II.
* Patients undergo squint surgery.

Exclusion Criteria:

* Declining to give written informed consent by patient legal guardian.
* Age younger than 3 years or older than 7 years.
* ASA classification ≥ III.
* History of allergy to the medications used in the study or egg products.
* Psychiatric disorder
* Other co-morbidities or congenital anomalies or neurological.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
the overall incidence of postoperative Emergence Agitation | EA incidence and severity will be determined using (PAED) scale at extubation (E0), upon arrival to the Post Anesthesia Care Unit (PACU) E1 and after 15 minute (E2), then after 30 minute in the PACU (E3).
  Pediatric Anesthesia Emergence Delirium (PAED) scale will be use to assess the incidence of Emergence Agitation (EA) A PAED score of 10 or higher is considered to be diagnostic of EA, but a score of 12 or higher is more sensitive and specific.

SECONDARY OUTCOMES:
heart rate changes | 30 minutes in the PACU
  heart rate (HR) will be measured at extubation , upon arrival to the PACU and after 15 minutes , then after 30 minutes in the PACU.
mean arterial pressure (MAP) changes | 30 minutes in the PACU
  mean arterial pressure (MAP) will be measured at extubation , upon arrival to the PACU and after 15 minutes , then after 30 minutes in the PACU.
peripheral oxygen saturation (SpO2) changes | 30 minutes in the PACU
  peripheral oxygen saturation (SpO2) will be measured at extubation , upon arrival to the PACU and after 15 minutes , then after 30 minutes in the PACU.
Proportion of patients with adverse events in the PACU | assessed up to 30 minutes after arrival of patient to PACU.
  including oxygen desaturation defined as SpO2 < 90%, regarded as severe desaturation when SpO2 < 85%, bradycardia defined as HR < 80 beats/min , shivering, dizziness, laryngospasm, severe coughing, and reintubation.
Proportion of patients with Post Operative Nausea and Vomiting (PONV) | assessed up to 30 minutes after arrival of patient to PACU.
  evaluated by a 4-point PONV Scale .
Time to discharge from the PACU. | 60 minutes
  the time the patients needs to be stable and discharge from the PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No